CLINICAL TRIAL: NCT04711785
Title: Assessment of the Possible Beneficial Effects of an Integrated Program of Multicomponent Physical Exercise Tutored at Home Through an Integrated Computer System. Cohort Study
Brief Title: Beneficial Effects of an Integrated Program of Multicomponent Physical Exercise. Cohort Study
Acronym: Ros-Ita
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No recruitment possibility
Sponsor: Hospital de la Ribera (Other)
Collaborators: University of Valencia (Other)
Responsible Party: Principal Investigator, Francisco Jose Tarazona-Santabalbina, MD, Ph D, Hospital de la Ribera
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRibera001-12012021
Record Dates: First submitted 2021-01-12; First posted 2021-01-15 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Frailty; Geriatric Syndromes; Functional Recovery
Keywords: older adults; frailty; geriatric assessment; geriatric syndromes; multicomponent exercise program
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: Cohort study
Masking Description: Cohort study no masking presented.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Multicomponent exercise program twice a week (2 hours per week) during six months
  Interventions: Behavioral: Multicomponent exercise program
- Control Goup (No Intervention): Usual routine.

INTERVENTIONS:
Behavioral: Multicomponent exercise program — The exposed group will carry out the following program of specific muscle strength and cardio physical activity aimed at reducing frailty.
  For 2.5 hours per week.
  Arms: Intervention

SUMMARY:
The study has been designed to analyze the possible positive effects of a multicomponent physical exercise program monitored with an integrated electronic device system in dwelling-community frailty older adults.

The study will assess changes in physical, nutritional, cognitive, and psychological aspects after program finishes at six months.

Information will be collected by researchers at baseline, monthly and after study finishes.

DETAILED DESCRIPTION:
The aging process is associated with physiological changes that determine a decrease in functional reserve and limit the ability to respond to external factors.

Likewise, aging is associated with a deterioration of the regulatory processes that maintain the functional integration of the different organs and systems. A direct consequence of this phenomenon is the atypical presentation of highly prevalent diseases in the elderly. This atypical presentation of diseases in the elderly is responsible for the so-called geriatric syndromes, considered as specific nosological entities with a high frequency of presentation in the elderly, being included within the prevention, diagnosis and treatment strategies of geriatric medicine.

These syndromes can generate greater morbidity and consequences, sometimes more serious than the disease that produces them. Its systematic detection should be included in the anamnesis of the clinical history of the elderly. Geriatric syndromes are a group of conditions usually caused by the conjunction of diseases with a high prevalence in the elderly and which are the frequent origin of functional or social disability in the population. They are the manifestation of many diseases, but they are also the beginning of many other problems that we must take into account from their detection to establish a good prevention of them.

The hypothesis of this work is that in frail and pre-frail older adults who participate in an integrated program of multicomponent physical exercise tutored by means of an app will improve their functional situation and reverse their diagnoses of pre and frailty.

ELIGIBILITY:
Inclusion Criteria:

* Frailty
* Informed consent signature

Exclusion Criteria:

* Life expectancy less than 6 months
* Acute Ischemic coronariopathy event during the last three months
* Active cancer treatment (chemoteraphy or radiotherapy) during the last three months
* Major surgery during the last six months

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Frailty reversion. | Six months
  Linda Fried's frailty criteria. Score 0 Fit, 1-2 Prefrail, 3 or over Frail
Intrinsic capacity | Six months
  ICOPE questionnaire score
Quality of life objective and subjective | Six months
  EuroQool 5 Dimensions (EQ-5D). Objective score 0 to 10.
Polypharmacy | Six months
  Quantitative definition. Considered polypharmacy the daily intake of 5 or more drugs.
Cognitive state | Six months
  Pfeiffer questionnaire
Depression | Six months
  Yesavage's Geriatrics Depression Scale (15 items)
Nutrition state | Six months
  Mini Nutritional Assessment Short Form. Score 0 to 14.
Falls | Six months
  Number of falls during follow-up period
Sarcopenia | Six months
  European Working Group on Sarcopenia in Older People (EWGSOP) criteria

SECONDARY OUTCOMES:
Hospital admissions | Six months
  Number of hospital admissions during follow-up period
Visits to General Practitioner (GP) | Six months
  Number of visits to GP during follow-up period
Validation of a shaking measurement tool to asses muscle strength | six months
  Gold standard Hand grip measured by dinamometry
Validation of a gait speed mobile phone tool | Six months
  Gold standard Gait speed measurement
Validation of a pulmonar capacity mobile phone tool | six months
  Gold standard forced expiratory volume in 1 (FEV1) Forced vital capacity (FVC)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco J Tarazona Santabalbina, MD, PhD, Principal Investigator — Hospital Universitario de la Ribera
Locations (1):
- Hospital Universitario de la Ribera, Alzira, Kingdom of Valéncia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martinez-Velilla N, Casas-Herrero A, Zambom-Ferraresi F, Saez de Asteasu ML, Lucia A, Galbete A, Garcia-Baztan A, Alonso-Renedo J, Gonzalez-Glaria B, Gonzalo-Lazaro M, Apezteguia Iraizoz I, Gutierrez-Valencia M, Rodriguez-Manas L, Izquierdo M. Effect of Exercise Intervention on Functional Decline in Very Elderly Patients During Acute Hospitalization: A Randomized Clinical Trial. JAMA Intern Med. 2019 Jan 1;179(1):28-36. doi: 10.1001/jamainternmed.2018.4869. PMID 30419096
- [Background] Gine-Garriga M, Roque-Figuls M, Coll-Planas L, Sitja-Rabert M, Salva A. Physical exercise interventions for improving performance-based measures of physical function in community-dwelling, frail older adults: a systematic review and meta-analysis. Arch Phys Med Rehabil. 2014 Apr;95(4):753-769.e3. doi: 10.1016/j.apmr.2013.11.007. Epub 2013 Nov 27. PMID 24291597
- [Background] Sanders LMJ, Hortobagyi T, la Bastide-van Gemert S, van der Zee EA, van Heuvelen MJG. Dose-response relationship between exercise and cognitive function in older adults with and without cognitive impairment: A systematic review and meta-analysis. PLoS One. 2019 Jan 10;14(1):e0210036. doi: 10.1371/journal.pone.0210036. eCollection 2019. PMID 30629631
- [Result] Tarazona-Santabalbina FJ, Gomez-Cabrera MC, Perez-Ros P, Martinez-Arnau FM, Cabo H, Tsaparas K, Salvador-Pascual A, Rodriguez-Manas L, Vina J. A Multicomponent Exercise Intervention that Reverses Frailty and Improves Cognition, Emotion, and Social Networking in the Community-Dwelling Frail Elderly: A Randomized Clinical Trial. J Am Med Dir Assoc. 2016 May 1;17(5):426-33. doi: 10.1016/j.jamda.2016.01.019. Epub 2016 Mar 3. PMID 26947059